CLINICAL TRIAL: NCT00123656
Title: Comparison of Esomeprazole to Aerosolized, Swallowed Fluticasone for Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: John C. Fang, M.D., University of Utah HSC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12790
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Esophagitis
Keywords: Eosinophilic esophagitis; esomeprazole; fluticasone
MeSH Terms: conditions — Esophagitis; Eosinophilic Esophagitis | interventions — Esomeprazole; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): fluticasone
  Interventions: Drug: fluticasone
- 2 (Active Comparator): esomeprazole
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: esomeprazole — esomeprazole dosed qam for 8 weeks
  Other Names: Nexium
  Arms: 2
Drug: fluticasone — fluticasone dosed 220 mcg 2 puffs swallowed BID for 8 weeks
  Other Names: Flovent
  Arms: 1

SUMMARY:
Eosinophilic esophagitis (EE) is a recently recognized entity. It has been thought to be related to both allergies and acid reflux. There have been reports that both swallowed, aerosolized steroids and proton pump inhibitors have been effective treatments. The researchers propose to directly compare the efficacy of aerosolized fluticasone to esomeprazole in the treatment of eosinophilic esophagitis. The hypothesis is that aerosolized fluticasone (Flovent) will be more effective in relieving symptoms of EE than esomeprazole (Nexium) treatment. Patients will undergo endoscopy, pH monitoring and manometry for diagnosis. Following diagnosis of EE by pathology (biopsy of esophagus), patients will be randomized to esomeprazole or swallowed fluticasone for 8 weeks. At the end of 8 weeks, subjects will be asked to repeat upper endoscopy with biopsies. Three questionnaires (dysphagia, gastroesophageal reflux disease [GERD], and allergy) will be completed by the patient at the first endoscopy and at the end endoscopy. The primary objective is to measure change in eosinophil infiltration of the esophagus in response to treatment of allergy (swallowed fluticasone) versus treatment for reflux (esomeprazole) in EE patients.

DETAILED DESCRIPTION:
This is a randomized, non-blinded, multicenter treatment trial to demonstrate and compare the efficacy of esomeprazole and fluticasone in the treatment of eosinophilic esophagitis.

Following the initial diagnostic EGD with four quadrant biopsy, serum eosinophil count and serum IgE levels will be measured. Patients will undergo 24 hour pH study to determine the incidence of reflux in this population. Clinical assessment will be performed with validated questionnaires quantifying dysphagia, GERD, and allergy/atopy. Patients will be randomized to 8 weeks of either esomeprazole versus swallowed aerosolized fluticasone. After 8 weeks of therapy, upper endoscopy will again be performed. Eosinophils per high power field will be quantified, and biopsies will be stained for major basic protein. Dysphagia, GERD, and allergy/atopy questionnaires will be repeated, as will serum eosinophil counts and IgE measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 with EE, defined as: a) dysphagia, food impaction or other upper gastrointestinal symptoms (chest pain, heartburn, regurgitation); b) multiple esophageal rings or furrows; c) the presence of >20 eosinophils/high power field in the squamous epithelium or deeper tissues of the esophagus
* Ability to undergo esophageal manometry and ambulatory pH monitoring
* No history of bleeding diathesis, significant cardiopulmonary disease, or other contraindication to upper endoscopy
* Those who have had a one month holiday from either esomeprazole therapy or fluticasone if they have been prescribed this prior to enrollment

Exclusion Criteria:

* Contraindication to proton pump inhibitors or swallowed fluticasone
* Need for immediate esophageal dilation at enrollment due to food impaction at the discretion of the performing endoscopist
* Inability to pass endoscope
* Pregnancy
* Incarceration
* Inability to provide informed consent
* History of esophago-gastric surgery or prior history of abdominal surgery with subsequent strictures or symptoms of obstruction such as abdominal pain and bloating
* Presence of other esophageal pathology that could account for patients' symptoms as determined by histological interpretation by the pathologist
* History of esophageal spasm resulting in trouble swallowing foods larger than 1 cm in diameter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To measure change in eosinophil infiltration and degranulation at 8 weeks in response to treatment of allergy versus treatment for GER in EE patients | 8 weeks

SECONDARY OUTCOMES:
To assess change in dysphagia score, GERD symptoms, allergy/atopy at 8 weeks using validated questionnaires | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John C. Fang, M.D., Principal Investigator — University of Utah HSC
Locations (1):
- University of Utah HSC, Salt Lake City, Utah, United States